CLINICAL TRIAL: NCT01507714
Title: Anterior Vaginal Wall Repair With Mesh in Combination With TVT-O to Reduce Urinary Stress Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0083-11EMC
Record Dates: First submitted 2012-01-02; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Preventive; tvt-o; stress incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control arm (No Intervention): vaginal wall repair surgery will be done to women in this arm, with no treatment for stress incontinence
- TVT-O arm (Active Comparator): the women in this arm will have a TVT-O procedure in addition to the vaginal wall repair
  Interventions: Procedure: Preventive transobturator tension free vaginal tape

INTERVENTIONS:
Procedure: Preventive transobturator tension free vaginal tape — during the vaginal wall repair surgery, a TVT-O procedure will be done
  Other Names: GYNECARE TVT™ Obturator System
  Arms: TVT-O arm

SUMMARY:
Urinary stress incontinence is defined as leakage of urine during stress. Urinary stress incontinence is a health problem with social, economic and psychological consequences. The appearance of Urinary stress incontinence post vaginal wall prolapse repair is a known phenomena. Part of the cases relate to pre-surgical occult Urinary stress incontinence which has been asymptomatic, and part of the cases relate to de-novo urinary stress incontinence post surgery. Latest studies have demonstrated 11-22% rate of post surgical urinary stress incontinence.

The aim of this study is to examine the efficacy of transobturator tension free vaginal tape (TVT-O) among women who intend to undergo vaginal wall repair by a vaginal approach.

DETAILED DESCRIPTION:
Urinary stress incontinence is defined as leakage of urine during stress (cough, lough, sneezing, coitus, heavy lifting, physical activity). Urinary stress incontinence is a health problem with social, economic and psychological consequences. The appearance of Urinary stress incontinence post vaginal wall prolapse repair is a known phenomena. Part of the cases relate to pre-surgical occult Urinary stress incontinence which has been asymptomatic, and part of the cases relate to de-novo urinary stress incontinence post surgery. Latest studies have demonstrated 11-22% rate of post surgical urinary stress incontinence.

The CARE study has examined the efficacy of preventive BURCH RETROPUBIC URETHROPEXY among women who underwent abdominal sacrocolpopexy. According to this study, the BURCH procedure reduced the rate of post surgery urinary stress incontinence. The authors recommend to offer those women the preventive surgery. Those results cannot be relied on when considering vaginal wall repair by the vaginal approach.

The aim of this study is to examine the efficacy of transobturator tension free vaginal tape (TVT-O) among women who intend to undergo vaginal wall repair by a vaginal approach.

ELIGIBILITY:
Inclusion Criteria:

* women with vaginal wall prolapse grade 2 and more
* no contraindication to vaginal wall repair or tvt-o
* No stress incontinence

Exclusion Criteria:

* urinary tract malformations
* past urinary stress incontinence surgical procedure
* UDI - question 17 or 18 - positive answer
* Occult urinary stress incontinence

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Stress incontinence | One year post operation
  The women will be classified as continent or not continent according to:
  * the Pelvic Floor Distress Inventory
  * stress test
  * need to other treatment for stress incontinence

SECONDARY OUTCOMES:
Surgical complications | one year
  Surgical complication
post surgery urgency or urge incontinence | one year
  urgency or urge incontinence

CONTACTS AND LOCATIONS:
Overall Officials: MEIRAV BRAVERMAN, MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- Dep of OG/GYN, Emek Medical Center, Afula, Israel